CLINICAL TRIAL: NCT06146725
Title: The RESBIOP-study: Resection Versus Biopsy in High-grade Glioma Patients (ENCRAM 2202)
Acronym: RESBIOP
Status: Recruiting | Type: Observational
Sponsor: Jasper Gerritsen (Other)
Collaborators: Haaglanden Medical Centre (Other); Universitaire Ziekenhuizen KU Leuven (Other); University Hospital Heidelberg (Other); Technical University of Munich (Other); Insel Gruppe AG, University Hospital Bern (Other); Massachusetts General Hospital (Other); University of California, San Francisco (Other)
Responsible Party: Sponsor-Investigator, Jasper Gerritsen, Jasper K.W. Gerritsen MD PhD, Erasmus Medical Center
Organization: Erasmus Medical Center (Other)
Other Study IDs: MEC-2020-0812-3
Record Dates: First submitted 2023-11-18; First posted 2023-11-27 (Actual); Last update posted 2023-11-27 (Actual); Status verified 2023-11

CONDITIONS: Glioblastoma; Glioblastoma, IDH-wildtype; Glioblastoma Multiforme; Glioblastoma Multiforme, Adult; Glioblastoma Multiforme of Brain
Keywords: Resection; Biopsy; Survival; Quality of life
MeSH Terms: conditions — Glioblastoma | interventions — Transurethral Resection of Bladder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Tumor resection: Tumor resection
  Interventions: Procedure: Tumor resection
- Tumor biopsy: Tumor biopsy
  Interventions: Procedure: Tumor biopsy

INTERVENTIONS:
Procedure: Tumor resection — Maximal safe resection of the tumor
  Groups: Tumor resection
Procedure: Tumor biopsy — Biopsy of the tumor
  Groups: Tumor biopsy

SUMMARY:
There are no guidelines or prospective studies defining the optimal surgical treatment for gliomas of older patients (≥70 years) or those with limited functioning performance at presentation (KPS ≤70). Therefore, the decision between resection and biopsy is varied, amongst neurosurgeons internationally and at times even within an instiutition. This study aims to compare the effects of maximal tumor resection versus tissue biopsy on survival, functional, neurological, and quality of life outcomes in these patient subgroups. Furthermore, it evaluates which modality would maximize the potential to undergo adjuvant treatment.

This study is an international, multicenter, prospective, 2-arm cohort study of observational nature. Consecutive HGG patients will be treated with resection or biopsy at a 3:1 ratio. Primary endpoints are: 1) overall survival (OS) and 2) proportion of patients that have received adjuvant treatment with chemotherapy and radiotherapy. Secondary endpoints are 1) proportion of patients with NIHSS (National Institute of Health Stroke Scale) deterioration at 6 weeks, 3 months and 6 months after surgery 2) progression-free survival (PFS); 3) quality of life at 6 weeks, 3 months and 6 months after surgery and 4) frequency and severity of Serious Adverse Events (SAEs). Total duration of the study is 5 years. Patient inclusion is 4 years, follow-up is 1 year.

DETAILED DESCRIPTION:
Trial design This is an international, multicenter, prospective, observational, 2-arm cohort study (registration: clinicaltrials.gov ID number TBA). Eligible patients are treated with either resection or biopsy with a 3:1 ratio with a sequential computer-generated random number as subject ID.

Study objectives The primary study objective is to evaluate safety and efficacy of resection versus biopsy in HGG patients as measured by overall survival (OS) and receipt of adjuvant treatment with chemotherapy and radiotherapy. Secondary study objectives are to evaluate postoperative neurological morbidity, progression-free survival (PFS), postoperative quality of life and SAEs after resection or biopsy as measured by NIHSS deteriration, tumor progression on MRI scans, quality of life questionnaires (QLQ C30, EORTC QLQ BN20, EQ 5D), and recording SAEs respectively.

Study setting and participants Patients will be recruited from the neurosurgical or neurological outpatient clinic or through referral from general hospitals of the participating neurosurgical hospitals, located in Europe and the United States. The study is carried out by centers from the ENCRAM Consortium.

Study patients are allocated to either the supramaximal or maximum safe resection group and will undergo evaluation at presentation (baseline) and during the follow-up period at 6 weeks, 3 months, 6 months and 12 months postoperatively. Motor function will be evaluated using the NIHSS (National Institute of Health Stroke Scale) scale. Cognitive function will be assessed using the Montreal Cognitive Assessment (MOCA). Patient functioning with be assessed with the Karnofsky Performance Scale (KPS) and the ASA (American Society of Anesthesiologists) physical status classification system. Health-related quality of life (HRQoL) will be assessed with the EORTC QLQ C30, EORTC QLQ BN20 and EQ 5D questionnaires. Overall survival and progression-free survival will be assessed at 12 months postoperatively. We expect to complete patient inclusion in 4 years. The estimated duration of the study (including follow-up) will be 5 years.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years and ≤90 years
2. Tumor diagnosed as HGG (WHO grade III/IV) on MRI as assessed by the neurosurgeon
3. Written informed consent

Exclusion Criteria:

1. Tumors of the cerebellum, brainstem or midline
2. Medical reasons precluding MRI (e.g. pacemaker)
3. Inability to give written informed consent
4. Secondary high-grade glioma due to malignant transformation from low-grade glioma
5. Second primary malignancy within the past 5 years with the exception of adequately treated in situ carcinoma of any organ or basal cell carcinoma of the skin

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with primary high-grade glioma will be recruited from the neurosurgical or neurological outpatient clinic or through referral from general hospitals of the participating neurosurgical hospitals, located in Europe and the United States. The study is carried out by centers from the ENCRAM Consortium.
Sampling Method: Non-Probability Sample
Enrollment: 564 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2028-01-01 (Estimated); Study Completion 2029-01-01 (Estimated)

PRIMARY OUTCOMES:
Overall survival | Up to 5 years postoperatively
  Time from diagnosis to death from any cause
Adjuvant treatment with chemotherapy and radiotherapy | 6 months postoperatively
  Proportion of patients that have received adjuvant treatment with chemotherapy and radiotherapy after surgery

SECONDARY OUTCOMES:
Progression-free survival | Up to 5 years postoperatively
  Time from diagnosis to disease progression (occurrence of a new tumor lesions with a volume greater than 0.175 cm3, or an increase in residual tumor volume of more than 25%) or death, whichever comes first
Neurological morbidity at 6 weeks | 6 weeks postoperatively
  NIHSS deterioration of 1 point or more at 6 weeks after surgery
Neurological morbidity at 3 months | 3 months postoperatively
  NIHSS deterioration of 1 point or more at 3 months after surgery
Neurological morbidity at 6 months | 6 months postoperatively
  NIHSS deterioration of 1 point or more at 6 months after surgery
Quality of life at 6 weeks (EORTC QLQ C30) | 6 weeks postoperatively
  Quality of life as assessed by the EORTC QLQ C30 questionnaire
Quality of life at 3 months (EORTC QLQ C30) | 3 months postoperatively
  Quality of life as assessed by the EORTC QLQ C30 questionnaire
Quality of life at 6 months (EORTC QLQ C30) | 6 months postoperatively
  Quality of life as assessed by the EORTC QLQ C30 questionnaire
Quality of life at 6 weeks (EORTC QLQ BN20) | 6 weeks postoperatively
  Quality of life as assessed by the EORTC QLQ BN20 questionnaire
Quality of life at 3 months (EORTC QLQ BN20) | 3 months postoperatively
  Quality of life as assessed by the EORTC QLQ BN20 questionnaire
Quality of life at 6 months (EORTC QLQ BN20) | 6 months postoperatively
  Quality of life as assessed by the EORTC QLQ BN20 questionnaire
Quality of life at 6 weeks (EQ-5D) | 6 weeks postoperatively
  Quality of life as assessed by the EQ-5D questionnaire
Quality of life at 3 months (EQ-5D) | 3 months postoperatively
  Quality of life as assessed by the EQ-5D questionnaire
Quality of life at 6 months (EQ-5D) | 6 months postoperatively
  Quality of life as assessed by the EQ-5D questionnaire
Serious Adverse Events | 6 weeks postoperatively
  Serious Adverse Events within 6 weeks postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Jasper Gerritsen, MD PhD, Principal Investigator — Erasmus Medical Center
Locations (8):
- United States (2):
  - University of California, San Francisco, San Francisco, California
  - Massachusetts General Hospital, Boston, Massachusetts
- University Hospital Leuven, Leuven, Belgium
- Germany (2):
  - Technical University Munich, Munich, Bavaria
  - University Hospital Heidelberg, Heidelberg
- Netherlands (2):
  - Erasmus Medical Center, Rotterdam, South Holland
  - Haaglanden Medical Center, The Hague
- Inselspital Universitätsspital Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Gerritsen JKW, Young JS, Krieg SM, Jungk C, Ille S, Schucht P, Nahed BV, Broekman MLD, Berger M, De Vleeschouwer S, Vincent AJPE. Resection versus biopsy in patients with glioblastoma (RESBIOP study): study protocol for an international multicentre prospective cohort study (ENCRAM 2202). BMJ Open. 2024 Sep 10;14(9):e081689. doi: 10.1136/bmjopen-2023-081689. PMID 39260848